CLINICAL TRIAL: NCT06123663
Title: A Study to Evaluate the Safety and Immunogenicity of a Single Dose of Adsorbed Tetanus Vaccine in a Population Aged 18 Years and Over
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-TTVA-001
Record Dates: First submitted 2023-11-01; First posted 2023-11-09 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2023-10

CONDITIONS: Tetanus
Keywords: Vaccine; Positive-controlled; Safety; ≥18 years
MeSH Terms: conditions — Tetanus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetanus Vaccine, Adsorbed (TTVA) (Experimental): 1 dose of (TTVA) (0.5ml)
  Interventions: Biological: TTVA
- Tetanus Vaccine, Adsorbed (TT) (Active Comparator): 1 dose of (TT) (0.5ml)
  Interventions: Biological: TT

INTERVENTIONS:
Biological: TTVA — Intramuscular injection, 1 dose of 0.5ml inoculated on Day 0
  Arms: Tetanus Vaccine, Adsorbed (TTVA)
Biological: TT — Intramuscular injection, 1 dose of 0.5ml inoculated on Day 0
  Arms: Tetanus Vaccine, Adsorbed (TT)

SUMMARY:
This is a randomized, observer-blind, positive-controlled study. There will be 2 treatment groups, Subjects who gave informed consent and passed the questioning screen were randomly assigned 1:1 to be immunized with 1 dose of Tetanus Vaccine, Adsorbed (TTVA) or control vaccine.

DETAILED DESCRIPTION:
Tetanus can be prevented with tetanus toxoid-containing vaccines (TT-containing vaccines, TTCVs), which are included globally in routine immunization programs for children, and in many countries at the time of prenatal care. China eliminated neonatal tetanus in 2012, but non-neonatal tetanus remains a serious public health problem. TT vaccine was first produced in 1924 and is used as a single antigen vaccine and combination vaccine component to prevent other vaccine-preventable diseases, including diphtheria, pertussis, poliomyelitis, hepatitis B, Haemophilus influenzae type b (Hib), and other vaccine-preventable diseases. Haemophilus influenzae type b (Hib)

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older, able to provide valid proof of identity for himself/herself.
* Ability to understand the requirements and process of the study and to agree to participate in the clinical trial and to sign an informed consent form.
* Ability to comply with the requirements of the clinical trial protocol and complete all follow-up studies.

Exclusion Criteria:

* Previously diagnosed tetanus infection.
* Vaccination against tetanus or vaccines containing tetanus toxoid antigen components (e.g., DPT, DPT, RCV, etc.) within 5 years.
* Axillary temperature >37.0°C on the day of enrollment.
* Women with a positive urine pregnancy test or during pregnancy or breastfeeding.
* Women of childbearing age, male volunteers and male volunteers whose partner is a woman of childbearing age have a pregnancy plan or birth plan during the study period.
* Persons suffering from thrombocytopenia, any coagulation disorder, or receiving anticoagulant therapy that may contraindicate intramuscular injection.
* Suffering from serious respiratory diseases, serious cardiovascular diseases, liver and kidney diseases, malignant tumors, serious infectious or allergic skin diseases, hypertension that cannot be controlled by medication (at the time of on-site measurement: systolic blood pressure ≥160mmHg, diastolic blood pressure ≥100mmHg), and being in the period of acute disease or chronic disease activity within 7 days.
* History of severe neurological disorders such as epilepsy, convulsions, encephalopathy, or history of psychiatric disorders.
* Previous history of severe allergy to vaccination or medication (anaphylaxis, anaphylactic laryngeal edema, anaphylactic purpura, thrombocytopenic purpura, localized anaphylactic necrotic reaction (Arthus reaction), etc.).
* Allergy to certain components of the vaccine used in this clinical trial (mainly tetanus toxoid, aluminum hydroxide, sodium chloride, etc.) or allergy to the above components from previous vaccination.
* Known or suspected immunological abnormalities (e.g., HIV infection, history of thyroid, pancreas, liver, spleen, kidney disease or resection), immunosuppressive therapy, cytotoxic therapy, systemic glucocorticosteroid medication (≥14 days) within 6 months prior to enrollment (excluding spray corticosteroid therapy for allergic rhinitis, surface corticosteroid therapy for acute uncomplicated dermatitis, etc.) topical medications).
* Received blood products (whole blood, component blood, immune globulin, etc.) in the previous 3 months or plan to use such products within 1 month of vaccination.
* Vaccination with live attenuated vaccine within 14 days, subunit vaccine or inactivated vaccine within 7 days.
* Plans to participate or is participating in clinical studies of any other drug.
* Abnormalities in preimmunization blood counts and blood biochemistry that are judged by the investigator to be clinically significant.
* Any circumstances that, in the judgment of the researcher, are likely to influence the assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions (AR) in subjects | 0-30 days after immunization

SECONDARY OUTCOMES:
Incidence of AR | 30 minutes after immunization
Incidence of adverse events (AE) | 0-30 days after immunization
Incidence of AR/AE | 0-7 days post-immunization
Proportion of laboratory safety indicators with clinically significant changes (CS), including hemoglobin level (HGB), white blood cell count (WBC), alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin (TBIL) | Day 8 post-immunization
Incidence of serious adverse events (SAEs) | 6 months post-immunization

CONTACTS AND LOCATIONS:
Overall Officials: Shiguang Lei, Principal Investigator — Guizhou Center for Disease Control and Prevention
Locations (1):
- Center for Disease Control and Prevention, Qixingguan District, Bijie City, Bijie, Guizhou, China